CLINICAL TRIAL: NCT02059421
Title: Comparative-effectiveness of Johrei Therapy and CBT-I in Facilitating Sleep in ICU Survivors
Brief Title: Johrei Therapy and CBT-I in Facilitating Sleep in ICU Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: The Johrei Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8674; The Johrei Institute (Other: Johrei Institute)
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disturbances in Survivors of Critical Illness
Keywords: Johrei therapy; Sleep; CBT-I; Critical illness
MeSH Terms: conditions — Critical Illness | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Johrei Therapy (Experimental): * 3 sessions per week lasting 30 minutes.
  * Daily report of bedtime and wake time.
  Baseline:
  * Polysomnography
  * Actigraphy
  * Questionnaires
  * Blood draw
  * Urine collection
    2 weeks:
  * Questionnaires
  * Actigraphy download
  * Sleep log reconciliation
    6 weeks:
  * Polysomnography
  * Actigraphy download
  * sleep log reconciliation
  * Questionnaires
  * Blood draw
  * Urine collection
  Interventions: Other: Johrei therapy
- Cognitive Behavioral Therapy for Insomnia (CBT-I) (Active Comparator): * 1 session per week for a total of 6 weeks with the option of 2 additional sessions.
  * Daily report of bedtime and wake time.
  Baseline:
  * Polysomnography
  * Actigraphy
  * Questionnaires
  * Blood draw
  * Urine collection
    2 weeks:
  * Questionnaires
  * Actigraphy download
  * Sleep log reconciliation
    6 weeks:
  * Polysomnography
  * Actigraphy download
  * sleep log reconciliation
  * Questionnaires
  * Blood draw
  * Urine collection
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — - Therapy session administered by a clinical psychologist using web-based video conferencing software.
  Therapy sessions will include:
  * Sleep restriction therapy
  * Stimulus control instructions
  * Sleep hygiene education
  Arms: Cognitive Behavioral Therapy for Insomnia (CBT-I)
Other: Johrei therapy — * Therapy will be administered by a senior Johrei administrator at the University of Arizona or the patient's residence.
  * Therapy sessions will consist of 3 sessions per week lasting 30 minutes each.
  * Therapist will wash his hands and and pray for 1 minute while facing the subject at a distance.
  * Therapy will be administered without physical contact.
  * During therapy the administrator will sit adjacent to the patient and channel energy from his palm towards the patient.
  Arms: Johrei Therapy

SUMMARY:
The purpose of this project is to compare the effectiveness of Johrei therapy (JT) and Cognitive-behavioral Therapy for Insomnia (CBT-I) in the treatment of sleep disturbances in survivors of critical illness. Subjects will be recruited following discharge from the Intensive Care Unit (ICU) and followed for 6 weeks. All subjects will undergo objective measurements of sleep quality and duration at baseline and at 6 weeks. Objective measurements will be made by portable (home-based) sleep studies and will wear a watch that measures sleep. Subjective measurements will be performed by sleep questionnaires: PSQI, Epworth sleepiness scale, sleep log, and Stanford Sleepiness Scale which will be performed at baseline, 2 and 6 weeks. A blood draw and urine collection will be done at both baseline and 6 weeks.

The central purpose of this proposal is to perform a comparative-effectiveness study of a complementary and alternative approach (Johrei therapy) and CBT-I in the treatment of sleep disturbances in survivors of critical illness. The investigators hypothesize that, in survivors of critical illness, Johrei therapy is superior or comparable to CBT-I in improving sleep quality (Pittsburgh Sleep Quality Index [PSQI] and sleep efficiency [measured by polysomnography]).

A secondary objective is to compare the effect of Johrei therapy and CBT-I on systemic markers of inflammation and urinary biomarkers of sleep and stress. The investigators hypothesize that, in survivors of critical illness, Johrei therapy is superior or comparable to CBT-I in reducing systemic markers of inflammation and urinary biomarkers of sleep and stress.

A tertiary objective is to determine whether the presence of insomnia or other sleep characteristics is associated with hospital readmissions within 30-days.

DETAILED DESCRIPTION:
Survivors of critical illness are known to have poor quality of life. Specifically, post-discharge insomnia symptoms were common and significantly associated with physical quality of life impairment among six-month acute lung injury (ALI) survivors, even after adjustment for post-traumatic stress disorder (PTSD) and depression symptoms. Further studies are needed to validate these results and to characterize sleep disturbance after ALI using sleep-specific metrics. Chronic insomnia impacts 1 in 10 adults and is linked to accidents, decreased quality of life, diminished work productivity, and increased long-term risk for medical and psychiatric diseases such as diabetes and depression. Insomnia and inadequate sleep is an under-recognized problem that ails the investigators society and nearly 8000 preventable deaths per year are attributed to fatigue-related motor vehicle crashes as compared to 13,000 attributable to drunken driving. In a National Gallup poll, it was estimated that nearly 70% of US residents do not get adequate sleep. Inadequate sleep has also been suggested to play a role in the causation and perpetuation of psychiatric disorders and has recently been labeled a carcinogen. Methods to improve sleep and vitality may decrease the effects of inadequate sleep and prevent diseases and deaths due to accidents. Moreover, sleep, or lack thereof, may be a reflection of global stress, disease severity, reveals much about patients' overall well-being and could be associated with hospital readmission.

Cognitive-behavioral therapy for insomnia (CBT-I) is currently considered the gold-standard treatment for insomnia. Recent National Institutes of Health consensus statements and the American Academy of Sleep Medicine's Practice Parameters recommend that cognitive-behavioral therapy for insomnia (CBT-I) be considered the first line treatment for chronic primary insomnia. Growing research also supports the extension of CBT-I for patients with persistent insomnia occurring within the context of medical and psychiatric co-morbidity. Sedative medications for insomnia may be associated with adverse side effects and have even been associated with all-cause mortality. Consequently, other non-pharmacological approaches have been gaining ground as therapeutic approaches for insomnia. Specifically, complementary and alternative forms of therapy such as yoga, mindful meditation, tai chi, Reikei and Johrei therapy have been used to promote sleep quality. Similar to Reikei, Johrei is a nondenominational spiritual practice and complementary and alternative medical therapy that channels the purification energy to a human body through the palm of its practitioner. Such an complementary and alternative treatment has previously been suggested to improve well-being and vitality in human studies. We know that well-being and vitality are facilitated by sleep and that sleep deprivation is associated with reduced well-being and vitality. Moreover, recently we showed that Johrei therapy improves sleep in a murine sleep deprivation model. Whether Johrei therapy achieves an improved sense of well-being through facilitation of sleep in survivors of critical illness is unknown. Specifically, whether or not Johrei therapy is comparable to CBT-I in the management of sleep problems in the survivors of critical illness is largely unknown. The proposed study will address this knowledge gap. If Johrei treatment can improve sleep in survivors of critical illness, patients with reduced vitality due to insufficient sleep (majority of US population), insomnia, and disrupted sleep (sleep apnea) may also benefit from such treatment.

Insomnia subjects, but not good sleepers, show high levels of pro-inflammatory cytokines that are associated with increased risk for heart disease and even mortality. Whether the improvement of sleep through CBT-I or Johrei therapy is mediated by reduction in stress and pro-inflammatory cytokine levels is unknown. The investigators study will address this knowledge gap by measuring circulating levels of cytokines in patients receiving Johrei therapy or CBT-I. Also, recent studies have shown that urinary levels of neurotransmitters may be increased (catecholamines such as epinephrine, norepinephrine, Ɣ-amino butyric acid (GABA)) or decreased (Taurine) in subjects with sleep disturbances. Whether or not CBT-I or other practices aimed at promoting sleep can normalize urinary changes in neurotransmitters is largely unknown.

A. JT arm: Johrei treatment will be administered to subjects at the University of Arizona or at the patient's residence for 3 sessions per week lasting 30 minutes each. Two of these sessions will be combined on one day with a 1 hour interval to yield two visits per week. A total of 18 sessions will be administered over the 6 weeks of participation. Therapy will be administered by a senior Johrei administrator who received his training from Reimei Kyokai in Kyoto, Japan. The Johrei will be administered as per all of the principles of Johrei. Before each therapy, the therapist will wash his hands and pray for 1 minute while facing the subject at a distance. The Johrei therapy will be administered without requiring physical contact by the placement of the therapist's hands in proximity of the subject (20 cms). Johrei therapy is a complementary and alternative form of therapy that originated in Japan, like Reiki therapy. Johrei therapy is a non-invasive bio-energy healing practice that is delivered by the outstretched hand of a Johrei practitioner (http://www.johrei-institute.org/aboutus.htm). Similar to Reiki, Johrei is a nondenominational spiritual practice and complementary and alternative medical therapy that channels the purification energy to a human body through the palm of its practitioner but without requiring physical touch. Such a complementary and alternative treatment has previously been suggested to improve well-being and vitality in human studies. We know that well-being and vitality are facilitated by sleep and that sleep deprivation is associated with reduced well-being and vitality. Moreover, recently we showed that Johrei therapy improves sleep in a murine sleep deprivation model.

B. CBT-I arm: Cognitive Behavioral therapy for Insomnia will be administered by a licensed and trained clinical psychologist after completion of initial assessment of the nature of the subjects sleep problems via a HIPAA-compliant encrypted Vsee app in the subject's iPAD. Weekly therapy will be administered in a manner that is tailored to suit the subject's need. A total of 6 sessions with an option of two additional sessions will be administered to help promote sleep. The administrator will go over techniques such as sleep restriction therapy, stimulus control instructions, and sleep hygiene education. Also, in order to prevent relapse, education will be provided regarding the extent to which they comprehend the patient's individual circumstances and critically reviewing the rules for good sleep, which in many instances need to be customized to each subject. All conversations and sessions with patients will take place in a manner designed to ensure privacy. For ensuring fidelity of the CBT-I sessions, 20% of the sessions will be video recorded at random for later review by clinical psychologist.

ELIGIBILITY:
Inclusion Criteria:

* Medical and surgical patients with recent critical illness warranting ICU stay.

Exclusion Criteria:

* Patients who are considered too unstable to undergo this investigation by their primary physician
* Patients with severe debilitating neurological disease ( end-stage Alzheimer's, large stroke, or other debilitating neurological disease) that renders patients incapable of providing informed consent
* Pregnancy (All inpatients with recent ICU stay of the childbearing age would have had a pregnancy test while in the hospital).
* Patient's residence is beyond a 20 mile radius from University of Arizona.
* Patient does not have a reliable way of communication such as a cellphone or telephone line.
* Being discharged to a nursing home of skilled nursing facility.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) (CBT-I, Johrei therapy) | 2 weeks
  Used to measure sleep quality
Polysomnography (CBT-I, Johrei therapy) | 6 weeks
  Used to measure sleep efficiency
Pittsburgh Sleep Quality Index (PSQI) (CBT-I, Johrei therapy) | 6 weeks
  Used to measure sleep quality.

SECONDARY OUTCOMES:
Actigraphy (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  Objectively measures periods of quiescence that could be inferred to be sleep.
Epworth Sleepiness Scale (ESS) (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  A measure of sleepiness
Sleep Log (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  Used to record bedtimes, wake times, and naps and will then be reconciled with actigraphy downloads.
Stanford Sleepiness Scale (SSS) (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  Measure of Alertness at different times during the day.
Post Traumatic Stress Disorder (PTSD) Checklist (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  Measures response to stressful life experiences.
PROMIS Sleep Related Impairment (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  Measures sleep impairment
PROMIS Sleep Disturbance (CBT-I, Johrei therapy) | Baseline, 2 weeks, 6 weeks
  Measures sleep disturbance
Rand 36 Item SF Health Survey Instrument (CBT-I, Johrei therapy) | 6 weeks
  Measures general health.
Cytokines and Neurotransmitters (CBT-I, Johrei therapy) | Baseline, 6 weeks
  Measures circulating levels of cytokines and neurotransmitters through blood and urine collection.

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD information.

REFERENCES:
- [Background] Buzzetti RA, Hinojosa-Kurtzberg M, Shea TJ, Ibuki Y, Sirakis G, Parthasarathy S. Effect of Johrei therapy on sleep in a murine model. Explore (NY). 2013 Mar-Apr;9(2):100-5. doi: 10.1016/j.explore.2012.12.004. PMID 23452712